CLINICAL TRIAL: NCT00005440
Title: Disability Among Adults With Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4369; R29HL048959 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-05

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To identify risk factors for work disability among adults with asthma treated by pulmonary and allergy specialists.

DETAILED DESCRIPTION:
BACKGROUND:

Disability among those with asthma is common and costly. Little is known about the causes of disability in asthma; experience with other chronic diseases suggests that illness severity alone does not adequately predict disability. There is a theoretical and experimental basis upon which to postulate that other variables, including factors such as job flexibility, asthma self-efficacy, social supports, and cigarette smoking may be predictors of disability in asthma. The study helped to explain the inter-relationships among illness severity, other co-factors and disability in asthma, addressing a major research gap.

DESIGN NARRATIVE:

The study was a cross-sectional survey, including retrospective work history data. A random sample was conducted of 40 board certified pulmonologists in Northern California enrolling persons with asthma. Pulmonologists maintained a log of all persons meeting a clinical definition of asthma presenting to their offices for treatment over a one month period. A total of 601 subjects with any history of laborforce participation were interviewed by a trained survey worker in order to assess severity of disease using a severity scale based on symptoms, medications, and past-asthma history. The computer-assisted, telephone-administered interviews used established survey instruments to assess psychosocial variables, smoking exposure and work history.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-09; Study Completion 1997-01 (Actual)

REFERENCES:
- [Background] Blanc PD, Cisternas M, Smith S, Yelin EH. Asthma, employment status, and disability among adults treated by pulmonary and allergy specialists. Chest. 1996 Mar;109(3):688-96. doi: 10.1378/chest.109.3.688. PMID 8617077
- [Background] Katz PP, Yelin EH, Smith S, Blanc PD. Perceived control of asthma: development and validation of a questionnaire. Am J Respir Crit Care Med. 1997 Feb;155(2):577-82. doi: 10.1164/ajrccm.155.2.9032197. (Retraction: PMID 10988083 Katz PP, Yelin EH, Blanc PD, Bainton DF. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):788)